CLINICAL TRIAL: NCT01205815
Title: Storage and Research Use of Human Bio-specimens From Melanoma Patients and Clinical Testing for Assignment of Treatment
Status: Recruiting | Type: Observational
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Responsible Party: Principal Investigator, Douglas Johnson, Associate Professor of Medicine, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC MEL 09109
Record Dates: First submitted 2010-09-17; First posted 2010-09-21 (Estimated); Last update posted 2025-09-19 (Actual); Status verified 2025-03

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Histocompatibility Testing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Tissue and blood collection — Tissue will be obtained from a previous biopsy if available, or if unavailable, tissue will be collected from a scheduled biopsy. About3-4 teaspoons of blood will be collected.

SUMMARY:
The purpose of this research is to identify biological characteristics occurring in the initiation and progression of melanoma.

ELIGIBILITY:
Inclusion criteria

* Pathologically-proven diagnosis of melanoma.
* Patient must have a test or procedure that has the potential to provide left-over tissue that can be banked for future research purposes OR the patient has already had a diagnostic or therapeutic procedure but who has not yet been approached to participate is also eligible.

Exclusion criteria

* Any patient with significant contraindications to venipuncture (e.g., severe anemia) will be excluded from blood collection procedures. However, if the patient provides consent and a paraffin-embedded block or 10-15 unstained slides of their tissue diagnosis, they will not be excluded from this protocol.
* Any patient unable or unwilling to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with melanoma.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2010-06-03 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Molecular changes in patients' melanoma tissue | at 120 months
  Tissue is collected upon consent or upon receipt of parafin block, primary aim will be met when all tissues are collected and analyzed at conclusion of study. Intent is to aid patients and their treating physician when making treatment decisions.

SECONDARY OUTCOMES:
Improve the time between ordering the test and results entry into medical records | 120 months
  To enhance the speed and detail of molecular mutation profiling of melanoma

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Johnson, M.D., Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbitl-Ingram Cancer Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Yan C, Saleh N, Yang J, Nebhan CA, Vilgelm AE, Reddy EP, Roland JT, Johnson DB, Chen SC, Shattuck-Brandt RL, Ayers GD, Richmond A. Novel induction of CD40 expression by tumor cells with RAS/RAF/PI3K pathway inhibition augments response to checkpoint blockade. Mol Cancer. 2021 Jun 6;20(1):85. doi: 10.1186/s12943-021-01366-y. PMID 34092233
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://www.vicc.org/ct/